CLINICAL TRIAL: NCT01465061
Title: A Survey on the Role and Benefits of Online Social Networks on Filipino Patients With Psoriasis
Status: Completed | Type: Observational
Sponsor: University of the Philippines (Other)
Collaborators: Philippine Dermatological Society (Network)
Responsible Party: Principal Investigator, Charlene U. Ang-Tiu, Dermatology resident, University of the Philippines
Other Study IDs: MED01032011
Record Dates: First submitted 2011-10-26; First posted 2011-11-04 (Estimated); Last update posted 2011-11-04 (Estimated); Status verified 2011-11

CONDITIONS: Psoriasis
Keywords: Online social network; Psoriasis; Filipino
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Online support user
  Interventions: Behavioral: Online support group

INTERVENTIONS:
Behavioral: Online support group — Joining online support group
  Other Names: Online social network, virtual online community

SUMMARY:
With the rise of usage of the internet, online social networks have recently been gaining popularity. Joining these groups can be beneficial to patients with chronic medical illness, such as psoriasis.This was a cross-sectional online survey of psoriasis patients in the Philippines who are members of online support groups. The survey was conducted for a period of three months.The purpose of the research project was to describe the demographics, disease characteristics, activities and benefits of online support groups to Filipino patients with psoriasis. The extent to which members experience empowering processes and outcomes was also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of psoriasis
* individuals who are willing to complete the online survey
* proficiency in English
* membership in an online psoriasis support network

Exclusion Criteria:

* nonmembers
* unwilling to participate in the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Members of virtual psoriasis local support networks (Yahoo-based Psoriasis Philippine Online Community, Inc. and Facebook Psoriasis Online Support Group) will be the main subjects of the study.
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2011-02; Primary Completion 2011-06 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Demographic profile of online support users | 3 months
  The sociodemographic profile of the respondents such as age (mean, range), sex, civil status, level of formal education, employment status were described.
Disease characteristics of online support users | 3 months
  The overall health status (poor, average, good), psoriasis severity (mild, moderate, severe), duration of illness of online support groups were evaluated.

SECONDARY OUTCOMES:
Activities performed and extent of participation of online support users | 3 months
  Participants were also asked regarding their attitudes and experiences with online communities, length of use, log-on frequency and nature of online activities.
Empowering processes and outcomes experienced by online support group members | 3 months
  The frequency with which empowering processes (exchange information, find recognition, share experiences, encounter emotional support, help others) occurred were measured on a 3-point scale (1-seldom to never, 2-sometimes, 3-often). The outcomes experienced (are better informed, feel more confident in relationship with physician, have improved acceptance, feel more confident with treatment, have enhanced social well-being, have increased optimism and control over the future, have enhanced self-esteem) were assessed on a 3-point scale (1-disagree, 2-neither agree nor disagree, 3-agree).
Correlation of variables | 3 months
  Intervariable correlation (overall health status/psoriasis severity with frequency/duration of usage, educational level/employment status with frequency of usage) were also be assessed for significance.

CONTACTS AND LOCATIONS:
Overall Officials: Charlene U Ang-Tiu, MD, Principal Investigator — University of the Philippines-Philippine General Hospital Section of Dermatology